CLINICAL TRIAL: NCT05212298
Title: Effects of Herbal Sleep Formula on Patients With Insomnia and Tinnitus: Prospective, Randomized, Double-blinded Clinical Trial
Brief Title: Effects of Herbal Sleep Formula on Patients With Insomnia and Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A10804001-4
Record Dates: First submitted 2021-08-27; First posted 2022-01-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disturbances; Tinnitus
MeSH Terms: conditions — Parasomnias; Tinnitus | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): receive placebo treatment, once a day, four pills each time.
  Interventions: Dietary Supplement: The gel contains a mixture of glucose and maltodextrin
- Herbal compound low-dose (Experimental): once a day, two herbal compound capsules and two placebos each time. The total amount of herbal compound capsules is 582 mg.
  Interventions: Dietary Supplement: Herbal compound low-dose
- Herbal compound high-dose (Experimental): once a day, four capsules each time. The total amount of herbal compound capsules is 1164 mg.
  Interventions: Dietary Supplement: Herbal compound high-dose

INTERVENTIONS:
Dietary Supplement: The gel contains a mixture of glucose and maltodextrin — The gel contains a mixture of glucose and maltodextrin - a complex carbohydrate - along with fat and a trace of protein.
  Arms: Control
Dietary Supplement: Herbal compound low-dose — The total amount of herbal compound capsules is 582 mg.
  Arms: Herbal compound low-dose
Dietary Supplement: Herbal compound high-dose — The total amount of herbal compound capsules is 1164 mg.
  Arms: Herbal compound high-dose

SUMMARY:
This project is planned to collect non-dialysis adults who suffer from sleep and tinnitus disorders and refuse to take sleeping medicines in our hospital by random assignment and double-blind method.

120 adults were divided into 3 groups.

1. Control group: receive placebo treatment, once a day, four pills each time.
2. Herbal compound low-dose group: once a day, two herbal compound capsules and two placebos each time. The total amount of herbal compound capsules is 582 mg.
3. Herbal compound high-dose group: once a day, four capsules each time. The total amount of herbal compound capsules is 1164 mg.

All subjects received health questionnaire, sleep questionnaire and tinnitus questionnaire before the start of the test At the end of the treatment(3 months), the health questionnaire, sleep questionnaire, and tinnitus questionnaire were accepted.

DETAILED DESCRIPTION:
Sleep disturbances were very popular in general population. The prevalence of sleep disturbances were about 20 ~30% in adults. Insomnia is a complex disease with many etiologies. For example, pressure from daily activity, psychiatric diseases, and organic diseases may contribute to sleep disturbances. Besides, insomnia often comorbid comorbidly with tinnitus, and form a vicious cycle between insomnia and tinnitus. In the aspect of treatment, besides psychological treatment, insomnia was often treated with hypnotics. Variable types of GABA agonists and/or antidepression agents, including selective serotonin reuptake inhibitor (SSRI) were often used for insomnia. However, the medical treatments for insomnia patients were unsatisfactory, and many patients search for traditional Chinese medicine and/or herbal medicine.

Tinnitus can be defined as a phantom auditory perception in the absence of an external sound source. It is a common auditory symptom with a prevalence ranges from 4.6% in a survey study in Iranian population to 25.3% in a nationally representative survey in the United States, depending on the definition of tinnitus and study populations. A recent nationwide survey of the general population of South Korea reported that the prevalence of any tinnitus was 20.7% among adults aged 20 to 98 years. The prevalence was higher in women and it increased with age. A cohort study in England indicated that the incidence of clinically significant tinnitus was 5.4 cases per 10,000 person-years.

Tinnitus can severely interfere with activities of daily living, with common comorbidities such as anxiety, irritability, depression, inability to concentration, and sleep disturbances. Studies based on both questionnaires and polysomnography reported that sleep disturbance are common in patients with tinnitus. Recently, the investigators found that the risk of tinnitus was increased in middle-aged and elderly patients with sleep disturbance and/or sleep apnea. In the aspect of treatment, GABA agonists were often used to for tinnitus, but the results are still unsatisfactory till now.

Since many years ago, traditional Chinese medicine or herbal medicine had take care of insomnia and tinnitus. Some herbal foods and/or drugs, for example Lemon Balm Extract、Rice bran fermentation extract (GABA)、L-Tryptophan, were suggested for these two diseases with various results. In this study ,the investigators aimed to investigate the effects of herbal sleep formula on the sleep and tinnitus of patients without hemodialysis or peritoneal dialysis.

This project is planned to collect non-dialysis adults who suffer from sleep and tinnitus disorders and refuse to take sleeping medicines in our hospital by random assignment and double-blind method.

120 adults were divided into 3 groups.

1. Control group: receive placebo treatment, once a day, four pills each time.
2. Herbal compound low-dose group: once a day, two herbal compound capsules and two placebos each time. The total amount of herbal compound capsules is 582 mg.
3. Herbal compound high-dose group: once a day, four capsules each time. The total amount of herbal compound capsules is 1164 mg.

All subjects received health questionnaire, sleep questionnaire and tinnitus questionnaire before the start of the test At the end of the treatment(3 months), the health questionnaire, sleep questionnaire, and tinnitus questionnaire were accepted.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20~70 years old
2. Non-dialysis patients
3. Suffering from sleep disorders and tinnitus
4. Refuse to take sleeping pills

Exclusion criteria:

1. Patients who are bedridden or unable to take care of themselves.
2. dialysis patients.
3. Patients who cannot understand the details of this study or cannot cooperate with the examination.
4. History of alcohol or drug abuse.
5. Pregnant and lactating women
6. Patients with moderate to severe sleep apnea
7. Take sleeping pills

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 3 month
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each aspect has a minimum score of 0 and a maximum of 3 points. The total score range is 0-21 points. When the PSQI score is greater than 5 points, it indicates that there is a sleep quality disorder. The higher the score, the worse the sleep quality.
Tinnitus Handicap Inventory | 3 month
  The Tinnitus Handicap Inventory (THI) comprises 25 items grouped into three subscales: Functional, Emotional, and Catastrophic. The Functional subscale (11 items) deals with limitations caused by tinnitus in the areas of mental, social, and physical functioning. The Emotional subscale (9 items) concerns affective responses to tinnitus, e.g. anger, frustration, depression, anxiety. The Catastrophic subscale (5 items) probes the most severe reactions to tinnitus, such as loss of control, inability to escape from tinnitus, and fear of having a terrible disease. For each item a patient can respond with a "yes" (scored 4 points), "sometimes" (2 points), or "no" (0 points). The responses are summed within each subscale and for the total scale. The higher the score, the greater the perceived tinnitus severity.

CONTACTS AND LOCATIONS:
Overall Officials: Juen-Haur Hwang, MD, PhD., Study Chair — Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City, Taiwan